CLINICAL TRIAL: NCT04155528
Title: The Effect of Music Therapy on Acute Pain and Sleep Quality Among Patients Underwent Abdominal Surgery: A Randomized Control Trial
Brief Title: Effect of Music Therapy on Postoperative Health Outcomes
Acronym: MToPOHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naglaa Fathy Afifi Youssef, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0163
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Music Therapy
Keywords: Music therapy; Pain; Sleep quality; Abdominal surgery
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): The intervention group will receive routine hospital care alongside 30 minutes of music therapy per day for three consecutive days. The music therapy will be initiated on the second day postoperatively. The assessment of baseline data and the music therapy will be applied at least three hours after analgesics administration.
  Interventions: Other: Music therapy
- Control group (No Intervention): Patients in the control group will receive routine hospital care only.

INTERVENTIONS:
Other: Music therapy — The intervention is listening to selected prerecorded music, specific Raga, on the individual CD player.
  Arms: Study group

SUMMARY:
Patients underwent surgical procedure experiences acute postoperative pain, but less than half report adequate postoperative pain relief. The poor management of pain after surgery is associated with inadequate sleep and poor mood. Music therapy is described as a non-pharmacological technique to accomplish individualized patient's goals for hospital treatment. Music has been used as a healing approach. In Saudi Arabia, there is a lack of evidence related to the effect of music therapy on pain and sleep among patients who underwent abdominal surgery. Studies are needed to address additional aspects of pain management and the promotion of sleep among Saudi adult postoperative people by using non-pharmacological modalities.

DETAILED DESCRIPTION:
Aim: The study will investigate the effect of music therapy on acute postoperative pain and sleep quality among patients undergoing abdominal surgery. A randomized control trial design will be demonstrated to accomplish this study. A total sample of 60 cases who underwent general abdominal surgery will be recruited. The study will be carried on in general surgery wards in one of a University Hospitals in Riyadh city, KSA. Four tools will be used to collect the data: Socio-demographic and medical data sheet, Pain Numeric Rating Scale (PNRS) for pain, Insomnia Severity Index (ISI) and Opinions Questions Regarding music therapy. The intervention group will listen to the selected prerecorded music on individual CD players by using a headset for consecutive three days. Music therapy will be given for 30 minutes during day time; depends upon the analgesics peak action time to avoid the bias of the intervention. Once again, it will be played before bedtime.

ELIGIBILITY:
Inclusion Criteria:

Patients who will meet the following criteria will be eligible to participate in this study:

* Adult patients, including both sexes and aged between18-60 years.
* Had an abdominal surgery.
* Give informed consent and are hemodynamically stabilized.
* Willing to receive music therapy for three consecutive postoperative days by using Headset.

Exclusion Criteria:

* Patients will be ineligible to participate in this study if they have any of the following:

  * Hearing deficit.
  * History of chronic pain.
  * Metastasis cancer, on narcotic medication.
  * Dementia, or psychiatric diagnosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-12-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (PNRS) | 3 days
  The Pain Visual Analogue Scale (VAS) is a standardized scale, which measures pain severity. The Pain Numeric Rating Scale (PNRS) is a numeric version of the VAS. The PNRS has a single 11-point numeric scale in which respondents select a number from 0 (no pain) to 10 (severe pain) that reflects their pain severity. The PNRS has a high test-retest reliability in both literate and illiterate patients (r = 0.96 & 0.95, respectively). Therefore, the PNRS will be used in this study to assess the pain severity.
Insomnia Severity Index (ISI) | 3 days
  The ISI is a widely used scale to evaluate insomnia. It consists of seven items; each item has a score of (0-4), where zero indicates no disturbance and four indicates very severe disturbance. The scale score gives four categories: no insomnia = 0-7; sub-threshold insomnia = 8-14; moderate insomnia = 15-21; and severe insomnia = 22-28. The Arabic ISI has ascertained satisfactory validity and reliability with a Cronbach's alpha coefficient of 0.84.

SECONDARY OUTCOMES:
Opinions Questions Regarding music therapy | 3 days
  This section has questions related to the participants' perspective regarding benefit in listening to music therapy during postoperative period in terms of reducing pain and improving sleep quality. There will be five questions which will evaluate the effect of music therapy in reducing pain and promoting sleep. This Question will be asked only to the participants in the experimental group at the end of the data collection. The questions are open ended or with dichotomous response (Yes or No). The results will be presented as percentage or frequency. There is no high or low answer, the score just reflects the participant's opinion on music as a therapy for reduce pain and improve sleep condition.

IPD SHARING:
Plan to Share IPD: No